CLINICAL TRIAL: NCT00601796
Title: Combination Immunotherapy for Lung Cancer
Brief Title: Vaccine Therapy, Tretinoin, and Cyclophosphamide in Treating Patients With Metastatic Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14744; P30CA076292 (NIH); NIH-OBA-0608-801 (Other: National Institute of Health)
Record Dates: First submitted 2008-01-19; First posted 2008-01-28 (Estimated); Results first posted 2013-05-15 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-02

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Cyclophosphamide; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Immunotherapy (Experimental): Vaccine + Cytoxan + ATRA as outlined in Detailed Description
  Interventions: Biological: Vaccine Treatment; Drug: Cyclophosphamide; Drug: All-trans retinoic acid (ATRA)

INTERVENTIONS:
Biological: Vaccine Treatment — We created a vaccine in which irradiated allogeneic lung adenocarcinoma cells are combined with a bystander K562 cell line transfected with hCD40L and hGM-CSF. By recruiting and activating dendritic cells, we hypothesized the vaccine would induce tumor regression in metastatic lung adenocarcinoma. Intradermal vaccine was given every 14 days x3, followed by monthly x3.
  Other Names: Allogeneic Tumor Cell-Based Vaccines
Drug: Cyclophosphamide — Cyclophosphamide (300 mg/m^2 IV) was administered before 1st and 4th vaccines to deplete regulatory T-cells.
  Other Names: cytoxan
Drug: All-trans retinoic acid (ATRA) — All-trans retinoic acid was given (150/mg/m^2/day) after 1st and 4th vaccines to enhance dendritic differentiation.
  Other Names: Vesanoid®; tretinoin; all trans retinoic acid; ATRA

SUMMARY:
The purpose of this study is to find out what effects (good and/or bad) a tumor vaccine used in combination with two drugs (ATRA and cytoxan) have on the patient and their cancer. We also want to find out if the vaccine and the drugs can boost the patient's immune system and how their immune system reacts, both before and after the vaccine treatment.

DETAILED DESCRIPTION:
This protocol describes a phase II study involving patients with stage IV adenocarcinoma of the lung. Treatment will consist of Cyclophosphamide (300 mg/m²) to be given IV on day 1 and day 57. On day 4 immunization with intradermal vaccine injections at 4 separate sites (bilateral upper arms and bilateral upper thighs will be repeated every 14 days times 2 followed by every 28 days times 3 (day 4, 18, 32, 60, 88, and 116). Decavac (tetanus shot) 0.5 cc intramuscular (IM) will be given after the first vaccine. ATRA (150 mg/m2/day) oral three times daily (TID) dosing administered after the first and fourth vaccines (day 5-7 & day 61-63). Those patients achieving stable disease (SD), partial response (PR), or complete response (CR) at restaging after the initial 6 vaccines will receive additional vaccines every 3 months until disease progression. The vaccine will consist of GM.CD40L bystander cells admixed with an equivalent number of the 2 allogeneic tumor cell lines. There will be a +/- 7 day window for all study related exams, tests, and procedures.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic adenocarcinoma of the lung
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, or 1
* No radiation therapy within 2 weeks of first vaccine administration
* No chemotherapy within 4 weeks of first vaccine administration
* No steroid therapy within 4 weeks of first vaccine administration
* Patient's written informed consent
* Adequate organ function (measured within a week of beginning treatment)
* Patients will be tested for human leukocyte antigen A0201 (HLA-A0201) as determined by flow cytometry followed by molecular analysis of a peripheral blood specimen, however this result will not be an inclusion criterion.
* Measurable metastatic tumor as defined by standard Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Lesions must be accurately measured in at least one dimension with the longest diameter greater than or equal 20mm. With spiral computer tomography (CT) scan, lesion must be greater than or equal to 10 mm at least one dimension.
* Patient's must have received, and completed first line chemotherapy.

Exclusion Criteria:

* Symptomatic brain metastasis
* Any acute medical problems requiring active intervention
* Current corticosteroid (other than replacement doses in patients who are hypoadrenal) or other immunosuppressive therapy
* Any other pre-existing immunodeficiency condition (including known HIV infection)
* Pregnant or lactating women -- Patients in reproductive age must agree to use contraceptive methods for the duration of the study (*A pregnancy test will be obtained before treatment).
* Eastern Cooperative Oncology Group (ECOG) performance status of 2, 3 or 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Chiappori, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 participants were accrued at a single center from 10/2006 to 6/2008.
Groups:
- Combination Immunotherapy: Vaccine + Cytoxan + ATRA as outlined in Detailed Description
  Vaccine Treatment : We created a vaccine in which irradiated allogeneic lung adenocarcinoma cells are combined with a bystander K562 cell line transfected with hCD40L and hGM-CSF. By recruiting and activating dendritic cells, we hypothesized the vaccine would induce tumor regression in metastatic lung adenocarcinoma. Intradermal vaccine was given every 14 days x3, followed by monthly x3.
  All-trans retinoic acid (ATRA) : All-trans retinoic acid was given (150/mg/m^2/day) after 1st and 4th vaccines to enhance dendritic differentiation.
  Cyclophosphamide : Cyclophosphamide (300 mg/m^2 IV) was administered before 1st and 4th vaccines to deplete regulatory T-cells.
Period: Overall Study
Arm/Group | Combination Immunotherapy
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 24 participants were accrued at a single center from 10/2006 to 6/2008. There were 14 participants with evaluable peripheral blood mononuclear cells (PBMCs).
Arm/Group | Combination Immunotherapy
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 12
Age Continuous [Median (Full Range); unit: years] | 64 [49 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Evaluable Participants With Tumor Response
Description: Number of participants with evaluable peripheral blood mononuclear cells (PBMCs) who demonstrated sustained tumor peptide-specific T-cell activation after vaccination. Peripheral blood mononuclear cells (PBMCs) were collected at baseline and after each vaccination. T-cell activation profiles were analyzed by ELISpot assay and tested by generalized Wilcoxon for correlation to survival.
Time Frame: 3 years
Population: 14 participants with evaluable PBMCs
Measure: Number; unit: participants
Arm/Group | Combination Immunotherapy
Number analyzed (Participants) | 14
participants | 5

2. Secondary Outcome: Median Time to Progression (TTP)
Description: Analysis of Time to Progression and Survival Endpoints. All patients will be considered in the analysis of progression free survival time (time from start of treatment to progression or death) and survival time (time from initiation of treatment to death). Progression is defined using the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
  Follow-up for this analysis will continue for all patients for their lifetimes. Time to progression and survival probabilities over time will be calculated by the method of Kaplan-Meier.
Time Frame: 3 years
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Immunotherapy
Number analyzed (Participants) | 24
months | 2.4 [0.3 to 4.6]

3. Secondary Outcome: Median Overall Survival (OS)
Description: Analysis of Time to Progression and Survival Endpoints. All patients will be considered in the analysis of progression free survival time (time from start of treatment to progression or death) and survival time (time from initiation of treatment to death). Follow-up for this analysis will continue for all patients for their lifetimes. Time to progression and survival probabilities over time will be calculated by the method of Kaplan-Meier.
Time Frame: 3 years
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Immunotherapy
Number analyzed (Participants) | 24
months | 8 [3.5 to 12.5]

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Toxicity will be assessed using the NCI Common Terminology Criteria for Adverse Criteria (CTAE-3),Version 3.0 (www.ctep.cancer.gov). Particular attention will assess the presence of symptomatic lymphadenopathy or any local skin / soft tissue reaction at the vaccine site. Blood tests for ANA and rheumatoid factor will be performed on any patient who develops evidence of autoimmune phenomena.
Time Frame: 3 years
Population: All participants
Measure: Number; unit: participants
Arm/Group | Combination Immunotherapy
Number analyzed (Participants) | 24
participants | 11

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Combination Immunotherapy
Serious Adverse Events (participants affected / at risk) | 11/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Immunotherapy (N=24)
Hemoglobin (Blood and lymphatic system disorders) | 1 (3)
Supraventricular and nodal arrhythmia - NOS (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (3)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (2)
Death not associated with CTCAE term - Disease progression - NOS (General disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (2)
Creatinine (Metabolism and nutrition disorders) | 1 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Abdomen - NOS (General disorders) | 1 (2)
Pain - Kidney (Renal and urinary disorders) | 1 (1)
Pain - Tumor pain (General disorders) | 2 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Obstruction, GU - Ureter (Renal and urinary disorders) | 1 (1)
Urine color change (Renal and urinary disorders) | 1 (1)
Vessel injury-vein - SVC (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Immunotherapy (N=24)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 19 (26)
Weight loss (General disorders) | 5 (5)
Insomnia (General disorders) | 4 (4)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 X 10^9/L) (General disorders) | 2 (2)
Rigors/chills (General disorders) | 2 (2)
Pain (General disorders) | 19 (44)
Pain - Head/headache (General disorders) | 14 (18)
Pain - joint (General disorders) | 6 (8)
Pain - back (General disorders) | 5 (5)
Pain - Abdomen - NOS (General disorders) | 3 (3)
Pain - Chest/thorax - NOS (General disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 10 (14)
Anorexia (Gastrointestinal disorders) | 9 (11)
Constipation (Gastrointestinal disorders) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (15)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 9 (9)
Alkaline phosphatase (Metabolism and nutrition disorders) | 6 (9)
Creatinine (Metabolism and nutrition disorders) | 6 (7)
Metabolic/Laboratory - other (Metabolism and nutrition disorders) | 3 (3)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 2 (2)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 8 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
Hemoglobin (Blood and lymphatic system disorders) | 9 (13)
Platelets (Blood and lymphatic system disorders) | 2 (3)
Allergic rhinitis (Immune system disorders) | 5 (5)
Allergy/Immunology - other (Immune system disorders) | 4 (4)
Mood alteration - Anxiety (General disorders) | 3 (4)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Hypertension (Cardiac disorders) | 3 (3)
Musculoskeletal/Soft - other (Musculoskeletal and connective tissue disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No